CLINICAL TRIAL: NCT06565299
Title: Cognitive and Speech Disorders in 5-7 Years Old Children With Congenital Heart Defects
Brief Title: Cognitive and Speech Disorders in Children With Congenital Heart Defects
Status: Completed | Type: Observational
Sponsor: Kemerovo State Medical University (Other)
Responsible Party: Principal Investigator, Evgeny Grigoryev, Head of the Department of Anesthesiology, Kemerovo State Medical University
Other Study IDs: 6
Record Dates: First submitted 2024-08-12; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cognition Disorder
Keywords: cognitive disoders; heart disease
MeSH Terms: conditions — Cognition Disorders; Heart Diseases | interventions — Cardiovascular Surgical Procedures; Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Children with family anamnesis confounding factorss, such as family composition, living conditions, conflict families (members of family suffering from any type of addiction, prisoned members of family, conflicts in front of a child's eyes).
  Interventions: Procedure: Cardiovascular surgery with cardiopulmonary bypass
- Group 2: without family anamnesis confounding factors
  Interventions: Procedure: Cardiovascular surgery with cardiopulmonary bypass

INTERVENTIONS:
Procedure: Cardiovascular surgery with cardiopulmonary bypass — Cardiovascular surgery about congenital heart defects with cardiopulmonary bypass

SUMMARY:
The study is aimed to found out expressive speech disorders as a sign of neurocognitive development delay in children with congenital heart defects before and after surgery

DETAILED DESCRIPTION:
The study will investigate the influence of congenital heart disease, operation and other health factors on neurocognitive and speech status of 5-7 years old children

ELIGIBILITY:
Inclusion Criteria:

* children with congenital heart disease that required total correction using cardiopulmonary bypass

Exclusion Criteria:

* patients with heart disease requiring palliative or endovascular correction, as well as children with chromosomal and genetic diseases (determined by karyotyping)

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 5-7 years old children with congenital heart defects bofore abd after cardiovascular operation with cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Neurocognitive status | 2 years
  Monitoring before the cardiovascular operation and in postoperative period (in 1 and 2 years).
  Assessment of speech disorders, short-term and long-term memory impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- Aleksandra Aeksandrovna Rumiantseva, Kemerovo, Kemerovo Oblast, Russia

IPD SHARING:
Plan to Share IPD: No